CLINICAL TRIAL: NCT00419484
Title: Effect of Pioglitazone on Cardiovascular Outcome on Higashi-Saitama Trial in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Dokkyo Medical University (Other)
Other Study IDs: 0309
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2007-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Type 2 Diabetes; Hypertension; Dyslipidemia; Diabetic Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Diabetic Nephropathies | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: pioglitazone

SUMMARY:
We want to investigate the effects of pioglitazone on cardiovascular events in Japanese patients with type 2 diabetes.

DETAILED DESCRIPTION:
Primary composite endpoints:

Cardiovascular death Non-fatal myocardial infarction and angina Non-fatal stroke Renal failure (hemodialysis/doubling of serum creatinine)

Secondary endpoints:

urinary albumin excretion diabetic retinopathy hyperlipidemia hypertension gout

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes HbA1c: more than 7% and less than 9%

Exclusion Criteria:

* insulin treatment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-03; Study Completion 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimasa Aso, MD, Principal Investigator — Dokkyo Medical University, Koshigaya Hospital
Locations (1):
- Dokkyo Medical University, Koshigaya Hospital, Koshigaya, Saitama, Japan